CLINICAL TRIAL: NCT07219472
Title: A Randomized, Single-Blind, Sham-Controlled Study of Scrambler Therapy for Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Scrambler Therapy for Chemotherapy-Induced Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: VelaSano (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE3Y25
Record Dates: First submitted 2025-10-20; First posted 2025-10-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; CIPN - Chemotherapy-Induced Peripheral Neuropathy
Keywords: Scrambler therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Scrambler Therapy (Experimental)
  Interventions: Device: Scrambler Therapy
- Sham Scrambler Therapy (Sham Comparator)
  Interventions: Other: Sham/No Intervention

INTERVENTIONS:
Device: Scrambler Therapy — Participants will attend 10 consecutive weekday 45-minute sessions of scrambler therapy.
  Arms: Scrambler Therapy
Other: Sham/No Intervention — Participants will be blinded as to which arm they are in (experimental vs. sham comparator), and as such, participants in the sham comparator arm will attend 10 consecutive weekday 45-minute sessions of sham scrambler therapy. In the sham comparator arm, participants will NOT receive a therapeutic level of scrambler therapy.
  Arms: Sham Scrambler Therapy

SUMMARY:
This research study is for people who have a condition called chemotherapy-induced peripheral neuropathy (CIPN). This condition develops as a result of receiving medication(s) to treat cancer, particularly chemotherapy. CIPN is characterized by pain, numbness, tingling or burning sensations, typically in the hands and feet of people. These symptoms can lead to physical suffering, limited ability to perform daily activities, and low quality of life. One of the ways to treat CIPN is using a device called Scrambler Therapy. Scrambler Therapy was approved by the Food and Drug Administration (FDA) in 2009 as a treatment for CIPN. The treatment involves electrical signals passing through wires attached to parts of the body via adhesive tabs near where symptoms of CIPN are experienced. A standard treatment course consists of 10 daily sessions lasting about one hour each. The purpose of this study is to determine the effect of a 10-day course of Scrambler Therapy on symptoms of chemotherapy-induced peripheral neuropathy, day-to-day activities, overall quality of life, and use of pain medications. Participants will be randomly assigned to one of two groups. One group will receive Scrambler Therapy. The other group will not receive it. Participants will not know which group they were in until after treatment has completed. Participants in the group who did not receive Scrambler Therapy will have the opportunity to receive it after one month. Participants will be in this research study about 12 to 14 months.

DETAILED DESCRIPTION:
Neuropathy is damage or disease affecting the somatosensory nervous system. It can result in pain, numbness and other feelings of tingling or burning on the skin. Neuropathic pain often does not go away for a long time, which can negatively impact quality of life. Even though neuropathic pain comes from the nervous system, it is often managed with medications.

In recent years, Scrambler Therapy (ST) has come up as a way to treat neuropathic pain that does not use medications. ST was approved by the FDA in 2009 to treat neuropathic pain. It works by replacing or overriding pain signals and rewires the way that people may perceive pain. It was originally designed to treat cancer pain. A standard course of ST consists of ten daily sessions over two consecutive weeks. Treatment may stop early if participants no longer report feeling neuropathic pain.

Previous research on the effects of ST for neuropathic pain have shown positive findings with very few participants reporting negative side effects of ST treatment. However, there are some limitations of ST, including the time and cost of the treatment, limited availability of ST, and the necessary skills needed to administer it.

ST is a promising solution to pain caused by CIPN. CIPN occurs in 30-40% of people treated with chemotherapy. CIPN can sometimes cause interruptions in cancer treatment and negatively impact quality of life. The amount of people with CIPN may also rise as more people with cancer live longer. Due to this, it is important to explore ST as a treatment for CIPN. This study aims to investigate the short-term and long-term impacts of ST as an alternative to medication treatments for CIPN.

ELIGIBILITY:
Inclusion Criteria:

* Adults with CIPN-related pain for at least three months duration, and for which the participant wants intervention
* At least three months from the last dose of neurotoxic cancer-directed drug
* No plan (at the time of study enrollment) for additional neurotoxic cancer-directed therapies for at least five months after trial enrollment
* Pain rated ≥ four out of 10 in severity (0-10 pain scale) during the seven days prior to enrollment
* > six-month life expectancy
* Able to complete questionnaires by themselves or with assistance
* Able to provide informed written consent
* ECOG Performance Status score ≥ two

Exclusion Criteria:

* Pregnant or nursing
* An operational implanted drug delivery system, implanted electronic medical device, life supporting medical device, and/or medical monitoring device
* History of myocardial infarction or ischemic heart disease within six months of trial enrollment
* History of epilepsy, brain damage resulting in seizure activity, or use of anticonvulsants for seizure
* Skin conditions such as open sores that will prevent proper application of electrodes
* Unwillingness or inability to wean and discontinue gabapentin or pregabalin prior to the start of ST
* History of symptomatic peripheral neuropathy prior to receiving neurotoxic chemotherapy
* Prior treatment with Scrambler Therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in participant-reported pain | Baseline, end of treatment (up to 14 days)
  Participant-reported pain is measured by the Severity of Neuropathic Symptoms, in which participants rank their pain on a scale of 0 (Not at All) to 10 (Severe). Higher scores indicate greater pain symptoms.

SECONDARY OUTCOMES:
Change in participant-reported non-pain neuropathic symptoms | Baseline, end of treatment (up to 14 days)
  Participant-reported non-pain neuropathic symptoms are measured by the Severity of Neuropathic Symptoms, in which participants rank their symptoms on a scale of 0 (Not at All) to 10 (Severe) for the following areas: numbness, tingling, cold sensation, warm sensation, stiffness, swelling, and pruritus. Higher scores indicate greater symptoms.
Change in functional status | Baseline, end of treatment (up to 14 days)
  Functional status is measured by the Functional Well-Being subscale of the Functional Assessment of Cancer Therapy - General (FACT-G) (version 4). This subscale contains 7 items, which participants will rank their functional status for each item on a 5-point scale of 0 (Not at all) to 4 (Very much). Lower scores indicate greater functional status.
Change in quality of life | Baseline, end of treatment (up to 14 days)
  Quality of life is measured by the Functional Assessment of Cancer Therapy - General (FACT-G) (version 4). It is a 27-item questionnaire with four subscales (physical well-being, social/family well-being, emotional well-being, and functional well-being). Participants answer questions on a 5-point scale from 0 (Not all all) to 4 (Very much). Lower scores indicate greater quality of life.
Change in participant-perceived treatment efficacy | Baseline, end of treatment (up to 14 days)
  Participant-perceived treatment efficacy is measured by the Patient Global Impression of Change, which is a single-item measure. Participants rank their belief about treatment efficacy on a 7-point scale from "Very much improved" to "Very much worse." Scores in the "improved" qualitative items indicate a greater perceived treatment efficacy.

OTHER OUTCOMES:
Change in participant-reported analgesic use for CIPN | Baseline, end of treatment (up to 14 days)
  Analgesic use will be measured by participant report of each type of and count of medication used in an attempt to lessen their neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Shoemaker, DO, MS, FAAHPM, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic
Locations (1):
- Case Comprehensive Cancer Center, Cleveland Clinic Foundation Taussig Cancer Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finnerup NB, Kuner R, Jensen TS. Neuropathic Pain: From Mechanisms to Treatment. Physiol Rev. 2021 Jan 1;101(1):259-301. doi: 10.1152/physrev.00045.2019. Epub 2020 Jun 25. PMID 32584191
- [Background] Szok D, Tajti J, Nyari A, Vecsei L. Therapeutic Approaches for Peripheral and Central Neuropathic Pain. Behav Neurol. 2019 Nov 21;2019:8685954. doi: 10.1155/2019/8685954. eCollection 2019. PMID 31871494
- [Background] Moisset X, Bouhassira D, Avez Couturier J, Alchaar H, Conradi S, Delmotte MH, Lanteri-Minet M, Lefaucheur JP, Mick G, Piano V, Pickering G, Piquet E, Regis C, Salvat E, Attal N. Pharmacological and non-pharmacological treatments for neuropathic pain: Systematic review and French recommendations. Rev Neurol (Paris). 2020 May;176(5):325-352. doi: 10.1016/j.neurol.2020.01.361. Epub 2020 Apr 7. PMID 32276788
- [Background] Marineo G. Inside the Scrambler Therapy, a Noninvasive Treatment of Chronic Neuropathic and Cancer Pain: From the Gate Control Theory to the Active Principle of Information. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419845143. doi: 10.1177/1534735419845143. PMID 31014125
- [Background] Majithia N, Smith TJ, Coyne PJ, Abdi S, Pachman DR, Lachance D, Shelerud R, Cheville A, Basford JR, Farley D, O'Neill C, Ruddy KJ, Sparadeo F, Beutler A, Loprinzi CL. Scrambler Therapy for the management of chronic pain. Support Care Cancer. 2016 Jun;24(6):2807-14. doi: 10.1007/s00520-016-3177-3. Epub 2016 Apr 4. PMID 27041741
- [Background] Wang EJ, Limerick G, D'Souza RS, Lobner K, Williams KA, Cohen SP, Smith TJ. Safety of Scrambler Therapy: A Systematic Review of Complications and Adverse Effects. Pain Med. 2023 Mar 1;24(3):325-340. doi: 10.1093/pm/pnac137. PMID 36069623
- [Background] Staff NP, Grisold A, Grisold W, Windebank AJ. Chemotherapy-induced peripheral neuropathy: A current review. Ann Neurol. 2017 Jun;81(6):772-781. doi: 10.1002/ana.24951. Epub 2017 Jun 5. PMID 28486769